CLINICAL TRIAL: NCT00948441
Title: Ethanol Lock Therapy for the Prevention of Catheter Related Blood Stream Infections
Brief Title: Pediatric Ethanol Lock Therapy Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Judy Martin, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08010189
Record Dates: First submitted 2009-07-07; First posted 2009-07-29 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Catheter-Related Infections
Keywords: intestinal insufficiency; central venous catheter; Catheter-Related Infections; pediatrics; ethanol
MeSH Terms: conditions — Catheter-Related Infections | interventions — Ethanol; Vascular Access Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): 25% ethanol for 12 weeks; wash out period for 4 weeks; heparin lock for 12 weeks
  Interventions: Drug: 25% ethanol; Other: heparin lock
- Group 2 (Experimental): heparin lock for 12 weeks; wash out period for 4 weeks; 25% ethanol lock for 12 weeks
  Interventions: Drug: 25% ethanol; Other: heparin lock

INTERVENTIONS:
Drug: 25% ethanol — Study Lock -25% Ethanol- The ethanol lock therapy consists of placing up to 2.3 ml of 25% ethanol into the central venous catheter and allowing it to dwell for 4 to 12 hours per day.
  Other Names: ethanol
Other: heparin lock — Placebo Lock - Heparin - These will be prepared in a sterile fashion in the Pharmacy of Children's Hospital of Pittsburgh in 10 day supplies as 1ml lock syringes utilizing 100 units/ml if the central venous catheter is accessed once daily and 10 units/ml if accessed more than once daily. The lock solution will be instilled and allowed to dwell for 4 to 12 hours.

SUMMARY:
This study is a double-blind crossover design to compare prophylaxis with ethanol lock therapy versus placebo lock therapy (heparin). The primary outcome measure will be the number of catheter related blood stream infections (CRBSI) in each time period.

DETAILED DESCRIPTION:
Central venous catheters (CVCs) are crucial for patients who require long term vascular access due to a variety of underlying diseases. Children with intestinal insufficiency and other diseases require vascular access to receive total parenteral nutrition, chemotherapy, fluid support and for the convenience of avoiding peripheral sticks when multiple blood draws are required. While these catheters have many benefits, they are also associated with complications such as catheter-related bloodstream infections (CRBSI). These infections can be a major cause of morbidity, mortality, and increased health care costs. Coagulase-negative staphylococci, Staphylococcus aureus, aerobic gram-negative bacilli, and Candida species (especially albicans) are the most common organisms responsible for these infections. These infections are traditionally treated with systemic antimicrobial therapy. There are times when the catheter must be removed to adequately treat the infection, however, indications for catheter removal in children are controversial. For some children with a history of multiple line infections, there are limited sites available to place new vascular access when the CVC needs to be replaced. Reducing the number of infections in this group of children is highly desirable. The goal of this study is to improve patient outcomes by reducing the risk of infection, thereby decreasing waitlist morbidity and mortality and improving post transplant care.

Lock therapy is the procedure of allowing medications to dwell in the line for extended periods of time without interruption. Many different agents such as ethanol, vancomycin and gentamicin have been used successfully as a means to salvage a CVC that has become infected. There is limited information regarding the use of lock therapy to prevent CRBSI in patients with CVCs. However, in patients with a history of multiple CRBSI, who have a critical need to maintain vascular access, lock therapy with a solution of 25% ethanol has been suggested to prevent future CRBSI. There is sufficient data to suggest that this combination is likely to be effective, is unlikely to lead to the development of multidrug resistant organisms and is well tolerated. Our hypothesis is that the use of ethanol as a lock therapy can reduce the number of CRBSI in both pre and post transplant patients with intestinal insufficiency.

Specific Aim: To compare the number of CRBSI in patients who receive ethanol lock therapy with the number of infections while on placebo lock therapy with heparin. This will be accomplished by conducting a prospective cross-over, double blind, placebo controlled study in children who have intestinal insufficiency and a history of multiple CRBSIs. Each child will receive 3 months of study lock therapy (25% ethanol) and 3 months of placebo lock therapy (heparin). The investigators, the patient and their family will be blinded to the treatment. The primary outcome measure will be the number of CRBSIs. Patients will also be observed for possible side effects from the therapy, and the need for line removal. This pilot study should provide preliminary data and information regarding the feasibility for a larger, multi-center study of ethanol lock therapy for the prevention of CRBSI.

ELIGIBILITY:
Inclusion criteria:

* patients with central venous access and a history of three or more CRBSI in the prior 6 months
* age greater than 6 months
* anticipation for the need for continued central venous access over the next 7 months
* availability to come for a monthly study visit
* anticipation that the patient will receive medical care at Children's Hospital of Pittsburgh for the majority of the CRBSI which occur during the next 7 months and the ability to lock the central venous catheter for a minimum of 4 hours per day

Exclusion criteria:

* age less than 6 months and greater than or equal to 21 years
* known immunodeficiency (with the exception of immunosuppression in a patient after organ transplantation)
* known allergy or intolerance to ethanol or heparin lock therapy

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith M Martin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children at our hospital with central venous access for parental nutrition and at least 3 CRBSI in the past 6 months were recruited. Patients had to be at least 6 months old and <21 years and be able to have a minimal dwell time of 4 hours. Exclusion criteria: known immunodeficiency or allergies to ethanol or heparin.
Pre-assignment Details: Randomized to one of two study groups. group 1 - ethanol lock followed by washout period followed by heparin lock. group 2 - heparin lock followed by washout period followed by ethanol lock.
Groups:
- 25% Ethanol/Washout/Heparin: First 25% ethanol, then Washout, then heparin
- Heparin Lock/Washout/25% Ethanol: First Heparin lock, then washout period, then 25% ethanol lock
Period: Overall Study
Arm/Group | 25% Ethanol/Washout/Heparin | Heparin Lock/Washout/25% Ethanol
Started | 8 | 8
Completed | 7 | 4
Not Completed | 1 | 4
Not completed — no longer meet inclusion criteria | 1 | 4

BASELINE CHARACTERISTICS:
Population: Children meeting the inclusion and exclusion criteria who received care at Children's Hospital of Pittsburgh were enrolled.
Groups:
- Group 1: 25% ethanol x12 weeks; washout x4 weeks; heparin x12 weeks
- Group 2: Heparin x12 weeks; washout x4 weeks; 25% ethanol x 12 weeks
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Full Range); unit: years] | 4.99 [1.2 to 13.5] | 2 [1.3 to 2.6] | 4 [1.2 to 13.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Episodes of Catheter Related Blood Stream Infections in Each Study Period.
Description: For the purpose of this study, episodes of catheter related blood stream infections were considered as the primary outcome measure. An episode of infection was defined as more than one positive blood culture obtained from the catheter requiring antibiotic therapy. Each episode after enrollment was recorded in its appropriate study period: ethanol lock, placebo lock, or washout period. If a patient had a catheter related blood stream infections, the study locks were held until after the number of days in each period was calculated as the number of days not on antibiotic therapy.
Time Frame: 7 months per study patient
Population: This was a crossover study. Each participant served as their own control. Infections in each time period of the study were compared. Infections with using ethanol locks and infections while using heparin locks.
Measure: Number; unit: number of CRBSI per 1000 catheter days
Groups:
- Infections While Using Ethanol Lock: 25% ethanol x 12 weeks
  25% ethanol: Study Lock -25% Ethanol- The ethanol lock therapy consists of placing up to 2.3 ml of 25% ethanol into the central venous catheter and allowing it to dwell for 4 to 12 hours per day.
- Infections While Using Heparin Lock: Heparin lock x 12 weeks
  heparin lock: Placebo Lock - Heparin - These will be prepared in a sterile fashion in the Pharmacy of Children's Hospital of Pittsburgh in 10 day supplies as 1ml lock syringes utilizing 100 units/ml if the central venous catheter is accessed once daily and 10 units/ml if accessed more than once daily. The lock solution was instilled and allowed to dwell for 4 to 12 hours.
Arm/Group | Infections While Using Ethanol Lock | Infections While Using Heparin Lock
Number analyzed (Participants) | 11 | 11
number of CRBSI per 1000 catheter days | 6.59 | 25.90
Statistical Analysis 1: Comparison: Infections While Using Ethanol Lock vs Infections While Using Heparin Lock; matched pairs T test to compare infection rates during the two study periods; Test type: Superiority or Other; p = 0.012, t-test, 2 sided

2. Secondary Outcome: Safety, Side Effects
Description: collection of adverse events and safety information. Each participant was contacted either at a clinical visit or by phone every two weeks while enrolled in the study.
Time Frame: 7 months per study patient
Population: collected adverse events during each time period
Measure: Number; unit: participants
Groups:
- Ethanol Lock: 25% ethanol
  25% ethanol: Study Lock -25% Ethanol- The ethanol lock therapy consists of placing up to 2.3 ml of 25% ethanol into the central venous catheter and allowing it to dwell for 4 to 12 hours per day.
- Heparin Lock: Heparin
  heparin lock: Placebo Lock - Heparin - These will be prepared in a sterile fashion in the Pharmacy of Children's Hospital of Pittsburgh in 10 day supplies as 1ml lock syringes utilizing 100 units/ml if the central venous catheter is accessed once daily and 10 units/ml if accessed more than once daily. The lock solution will be instilled and allowed to dwell for 4 to 12 hours.
Arm/Group | Ethanol Lock | Heparin Lock
Number analyzed (Participants) | 11 | 11
participants | 11 | 11

ADVERSE EVENTS:
Time Frame: 7 months during study participation
Description: Patients were seen in person (during hospitalization or clinic visit) or contacted by telephone every two weeks during the study enrollment period. Medical records were reviewed for adverse events.
Arm/Group | Ethanol Lock | Heparin Lock
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No